CLINICAL TRIAL: NCT03092271
Title: Randomized Trial of Stepped Care for Suicide Prevention in Teens and Young Adults
Acronym: Step2Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Kaiser Foundation Research Institute (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Joan Asarnow, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 112147; 16-001594 (Other: UCLA IRB)
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Suicidal Behavior; Self-Harm, Deliberate; Suicidal Ideation; Suicide
Keywords: suicide; suicide attempt; self harm; depression
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Suicide; Suicide, Attempted; Depression

STUDY DESIGN:
Intervention Model Description: Randomization to one of two conditions: 1) Zero suicide Best Practices/Quality Improvement; or 2) Zero suicide Best Practices/Quality Improvement plus stepped care for suicide prevention intervention
Who Masked: Outcomes Assessor
Masking Description: Assessments will be conducted by assessors who are naive to randomization assignment. Every effort will be made to conceal all information regarding randomization and randomization assignment to staff involved in assessment, recruitment, or other study activities that could lead to bias. It is not possible to conceal randomization status from intervention staff, as they will be delivering the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero Suicide Quality Improvement (ZSQI) (Active Comparator): Zero suicide best practices as implemented through a health system zero suicide quality improvement initiative
  Interventions: Behavioral: Zero Suicide Quality Improvement
- Stepped Care for Suicide Prevention (Experimental): ZSQI plus a stepped care intervention that matches intensity of services to youth risk level.
  Interventions: Behavioral: Stepped Care for Suicide Prevention; Behavioral: Zero Suicide Quality Improvement

INTERVENTIONS:
Behavioral: Stepped Care for Suicide Prevention — ZSQI plus Stepped Care for Suicide Prevention
  Arms: Stepped Care for Suicide Prevention
Behavioral: Zero Suicide Quality Improvement — ZSQI

SUMMARY:
This randomized controlled trial will evaluate two approaches to achieving the aspirational goal of Zero Suicide within a health system: 1) Zero Suicide Best Practices initiated through a zero suicide quality improvement initiative within a health system; and 2) Zero Suicide Best Practices plus an innovative stepped care for suicide prevention intervention for adolescents and young adults that matches treatment intensity with risk levels for suicide/self-harm. ..

DETAILED DESCRIPTION:
We propose a rigorous randomized trial to evaluate an innovative stepped care for suicide prevention intervention for adolescents and young adults, compared to a zero suicide program initiated by a health system. An effective zero suicide strategy for this age group is critically needed because this is a developmental period when: 1) suicide is the second leading cause of death, accounting for more deaths than any medical illness; 2) suicidal tendencies and behaviors often first occur in this age span; 3) rates of suicide and suicide attempts increase dramatically; and 4) effective intervention can reduce risk, suffering, and costs over lifetimes.

The project combines a partnership with a health system that has strong infrastructure and commitment to quality improvement for zero suicide with a research team that has successfully implemented collaborative stepped care interventions in health systems and has expertise in clinical, health services, economics, and policy research and dissemination. We will identify and enroll 300 youths ages 12-24 with elevated suicide and suicide attempt risk using a multi-stage screening process. Eligible youths will be randomized to: 1) zero suicide best practices, which emphasizes health system quality improvement (ZSQI); or 2) ZSQI plus stepped care for suicide prevention, which integrates evidence-based suicide prevention with primary care and emergency services. Prior research demonstrates the value of similar integrated medical-behavioral health interventions for improving patient outcomes, rates of care, and continuity of care- a critical issue for zero suicide efforts, as many youths discontinue care prematurely despite continuing risk. The ZSQI plus stepped care for suicide prevention approach uses: 1) risk assessments to triage youths to appropriate care levels; 2) care managers to deliver cognitive behavior therapy and dialectical behavior therapy skills training and support primary care and emergency clinicians with patient evaluation and treatment; 3) internet-delivered cognitive-behavior therapy and dialectical behavior therapy treatment components plus access to coaching support for lower risk youths, with stepped up in-person group and/or individual treatment added for higher risk youths; and 4) regular monitoring of patient outcomes, with feedback to clinicians to facilitate decision-making and use of the stepped care algorithms. The intervention period is 12 months: 6 months of acute treatment; and 6 months of continuation treatment. Results will provide critical information for health systems and science regarding the potential to achieve zero suicide goals by integrating state of the art science with practice quality improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Presence during past year of a suicide attempt, interrupted suicide attempt, aborted suicide attempt, or active suicidal ideation with a plan; or 2) past year depression, plus a history of a suicide attempt and/or recurrent self-harm;
2. Age 12-24 years

Exclusion Criteria:

1. Mental health/behavioral symptoms that would preclude productive engagement in study assessments or intervention (e.g., active psychosis; drug dependence)
2. Life threatening medical illness or other characteristics that would impede study participation (e.g. plans to move from Oregon during study period; plans for placement out of the home, insufficient locator information for follow-up)
3. Youth receives majority of mental health care outside of the Kaiser-Permanente health system.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 301 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Suicide Attempt Behavior | 12-month observation period
  fatal and nonfatal suicide attempts/suicide attempt behaviors

SECONDARY OUTCOMES:
Suicide Events | 12-month observation period
  fatal and nonfatal suicide attempts/suicide attempt behaviors, planning/preparatory acts, active suicidal ideation
Self Harm Episodes | 12-month observation period
  suicide attempts, undetermined self-harm, and nonsuicidal self-injury
Suicidality | 12-month observation period
  Continuous measure of suicidality
Depression | 12-month observation period
  Continuous depressive symptom score

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Kaiser Permanente Northwest, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No
Only fully anonymized and de-identified data as approved by the Institutional Review Board. The study principal investigator will collaborate with National Institute of Mental Health to finalize public use dataset procedures, ensure that the rights and privacy of all individual research participants are protected, and that Protected Personal Health Information is protected as required by law and approved by the study Institutional Review Board. The plan is for a limited access database of anonymized and de-identified data to be created. This data set will be available after study papers are completed and accepted for publication.

REFERENCES:
- [Derived] Asarnow JR, Clarke GN, Firemark AJ, Bedics J, Miranda J, Zhang L, Duan N, Comulada WS. Stratified Stepped-Care for Reducing Suicide Attempts and Self-Harm in Youth: A Randomized Clinical Trial. J Am Acad Child Adolesc Psychiatry. 2025 Dec 23:S0890-8567(25)02238-5. doi: 10.1016/j.jaac.2025.12.008. Online ahead of print. PMID 41448486
- [Derived] Sheppler CR, Edelmann AC, Firemark AJ, Sugar CA, Lynch FL, Dickerson JF, Miranda JM, Clarke GN, Asarnow JR. Stepped care for suicide prevention in teens and young adults: Design and methods of a randomized controlled trial. Contemp Clin Trials. 2022 Dec;123:106959. doi: 10.1016/j.cct.2022.106959. Epub 2022 Oct 11. PMID 36228984
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793